CLINICAL TRIAL: NCT07287046
Title: A Comparison of Efficacy Between High-intensity Laser Therapy and Focused Extracorporeal Shock Wave Therapy in Patient With Plantar Fasciitis; Single Blinded Randomize Controlled Study
Brief Title: A Single-Blind Randomized Controlled Study Comparing the Efficacy of High-Intensity Laser Therapy and Focused Extracorporeal Shock Wave Therapy in Patients With Plantar Fasciitis
Acronym: HILT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MURA2025/885; Ramathibodi Hospital (Other: Ramathibodi Hospital)
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HILT group (Experimental): High-power laser therapy (iLUX® XP) was applied using a power output of 6 W, an energy density of 5 J/cm², and a spot size of 10 cm², delivering a total energy of 150 J per session. Treatment consisted of 6 sessions, administered twice per week for 3 weeks.
  Interventions: Device: High power Laser therapy
- fESWT group (Active Comparator): Focused extracorporeal shock wave therapy (fESWT) using the DUOLITH® SD1 (STORZ Medical) was applied at a frequency of 4 Hz, starting at an energy flux density of 0.2 mJ/mm² and gradually increased as tolerated. Each session consisted of 2,000 shocks, for a total of 3 sessions (one session per week)
  Interventions: Device: Focused extracorporeal shock wave therapy

INTERVENTIONS:
Device: High power Laser therapy — High-power laser therapy (iLUX® XP) was applied using a power output of 6 W, an energy density of 5 J/cm², and a spot size of 10 cm², delivering a total energy of 150 J per session. Treatment consisted of 6 sessions, administered twice per week for 3 weeks
  Arms: HILT group
Device: Focused extracorporeal shock wave therapy — Focused extracorporeal shock wave therapy (fESWT) using the DUOLITH® SD1 (STORZ Medical) was applied at a frequency of 4 Hz, starting at an energy flux density of 0.2 mJ/mm² and gradually increased as tolerated. Each session consisted of 2,000 shocks, for a total of 3 sessions (one session per week)
  Arms: fESWT group

SUMMARY:
This randomized controlled trial aims to evaluate the efficacy of High-Intensity Laser Therapy (HILT) and Focused Extracorporeal Shock Wave Therapy (fESWT) in reducing pain in patients with plantar fasciitis. The study also examines the effects of HILT and fESWT on health-related outcomes, including VAS-FA, FFI, plantar fascia thickness, and adverse events.

Researchers will compare HILT with fESWT as treatment options for patients with plantar fasciitis.

Participants will receive either HILT or fESWT along with an exercise program. They will attend follow-up visits to assess outcomes at 1, 2, 3, 6, and 12 weeks after the first treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 years
* Pain was worse in the initial step after and an extended period of rest
* Pain was decreased initially after the first steps but exacerbated with increased activity
* VAS ≥ 4
* Pain was localized and sharp but not radiating,
* Pain was reproduced with palpation of the plantar fascia

Exclusion Criteria:

* Have Wound/Infection/tumor in treatment area
* History of foot trauma in 3 months
* History of intervention at plantar fascia in 6 months such as Ultrasound therapy, steroid injection, surgery or botulinum toxin injection
* Pain medication within one week before participation
* Patient wasn't desired to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-12-25 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | Pre-treatment, and at 1-, 2-, 3-, 6-, and 12-week post-treatment
  a pain rating scale based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale "no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm) Measurements from the starting point (left end) of the scale to the patients' marks are recorded in centimeters and are interpreted as their pain

SECONDARY OUTCOMES:
VAS-FA Thai version | Pre-treatment, and at 1-, 2-, 3-, 6-, and 12-week post-treatment
  The parameter used to assess the level of pain in several foot activities
Foot function index Thai version | Pre-treatment, and at 1-, 2-, 3-, 6-, and 12-week post-treatment
  a self-reporting questionnaire covering several dimensions of foot function categorized in 3 subscales that quantify the impacts of foot problems on pain, disability and activity limitation. FFI use a horizontal numeric block rating scale with 10 equal size boxes ranging from 0 to 9.
Thickness of plantar fasciitis | Pre-treatment, and 12-week post-treatment
  The plantar fascia thickness was measured at the point of plantar fascial insertion into the calcaneus with ultrasound machine in longitudinal view of tendon in both affected and healthy feet (mm). The quantitative measurement was achieved by recording the thickest part measured.
Adverse events | Pre-treatment, and at 1-, 2-, 3-, 6-, and 12-week post-treatment
  Including post-treatment soreness, burns, a burning sensation, and hematoma

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. Data will be analyzed and reported only in aggregate form in scientific publications, including baseline characteristics and study outcomes

REFERENCES:
- [Result] Sahni K, Sanyal B, Agrawal MS, Pant GC, Khanna NN, Khanna S. Carcinoma of breast associated with pregnancy and lactation. J Surg Oncol. 1981;16(2):167-73. doi: 10.1002/jso.2930160208. PMID 7464155
- [Result] Morrissey D, Cotchett M, Said J'Bari A, Prior T, Griffiths IB, Rathleff MS, Gulle H, Vicenzino B, Barton CJ. Management of plantar heel pain: a best practice guide informed by a systematic review, expert clinical reasoning and patient values. Br J Sports Med. 2021 Oct;55(19):1106-1118. doi: 10.1136/bjsports-2019-101970. Epub 2021 Mar 30. PMID 33785535
- [Result] Alam M, Warycha M. Complications of lasers and light treatments. Dermatol Ther. 2011 Nov-Dec;24(6):571-80. doi: 10.1111/j.1529-8019.2012.01476.x. PMID 22515672
- [Result] Ermutlu C, Aksakal M, Gumustas A, Ozkaya G, Kovalak E, Ozkan Y. Thickness of plantar fascia is not predictive of functional outcome in plantar fasciitis treatment. Acta Orthop Traumatol Turc. 2018 Nov;52(6):442-446. doi: 10.1016/j.aott.2018.01.002. Epub 2018 Oct 9. PMID 30314878
- [Result] Angthong C, Chernchujit B, Suntharapa T, Harnroongroj T. Visual analogue scale foot and ankle: validity and reliability of Thai version of the new outcome score in subjective form. J Med Assoc Thai. 2011 Aug;94(8):952-7. PMID 21863677
- [Result] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Result] Keskula DR, Tamburello M. Conservative management of piriformis syndrome. J Athl Train. 1992;27(2):102-10. PMID 16558144
- [Result] Naruseviciute D, Kubilius R. The effect of high-intensity versus low-level laser therapy in the management of plantar fasciitis: randomized participant blind controlled trial. Clin Rehabil. 2020 Aug;34(8):1072-1082. doi: 10.1177/0269215520929073. Epub 2020 Jun 8. PMID 32513018
- [Result] Gollwitzer H, Diehl P, von Korff A, Rahlfs VW, Gerdesmeyer L. Extracorporeal shock wave therapy for chronic painful heel syndrome: a prospective, double blind, randomized trial assessing the efficacy of a new electromagnetic shock wave device. J Foot Ankle Surg. 2007 Sep-Oct;46(5):348-57. doi: 10.1053/j.jfas.2007.05.011. PMID 17761319
- [Result] Huffer D, Hing W, Newton R, Clair M. Strength training for plantar fasciitis and the intrinsic foot musculature: A systematic review. Phys Ther Sport. 2017 Mar;24:44-52. doi: 10.1016/j.ptsp.2016.08.008. Epub 2016 Aug 18. PMID 27692740
- [Result] Porter D, Barrill E, Oneacre K, May BD. The effects of duration and frequency of Achilles tendon stretching on dorsiflexion and outcome in painful heel syndrome: a randomized, blinded, control study. Foot Ankle Int. 2002 Jul;23(7):619-24. doi: 10.1177/107110070202300706. PMID 12146772
- [Result] Petraglia F, Ramazzina I, Costantino C. Plantar fasciitis in athletes: diagnostic and treatment strategies. A systematic review. Muscles Ligaments Tendons J. 2017 May 10;7(1):107-118. doi: 10.11138/mltj/2017.7.1.107. eCollection 2017 Jan-Mar. PMID 28717618
- [Result] Zare Bidoki M, Vafaeei Nasab MR, Khatibi Aghda A. Comparison of High-intensity Laser Therapy with Extracorporeal Shock Wave Therapy in the Treatment of Patients with Plantar Fasciitis: A Double-blind Randomized Clinical Trial. Iran J Med Sci. 2024 Mar 1;49(3):147-155. doi: 10.30476/IJMS.2023.98042.2991. eCollection 2024 Mar. PMID 38584653
- [Result] Thammajaree C, Theapthong M, Palee P, Pakpakorn P, Sitti T, Sakulsriprasert P, Bunprajun T, Thong-On S. Effects of radial extracorporeal shockwave therapy versus high intensity laser therapy in individuals with plantar fasciitis: A randomised clinical trial. Lasers Med Sci. 2023 May 23;38(1):127. doi: 10.1007/s10103-023-03791-5. PMID 37219650
- [Result] Ordahan B, Karahan AY, Kaydok E. The effect of high-intensity versus low-level laser therapy in the management of plantar fasciitis: a randomized clinical trial. Lasers Med Sci. 2018 Aug;33(6):1363-1369. doi: 10.1007/s10103-018-2497-6. Epub 2018 Apr 7. PMID 29627888
- [Result] Ebid AA, Alhammad RM, Alhendi RT, Alqarhi BA, Baweyan EM, Alfadli LH, Alzahrani MA, Alotaibi MF, Alaidrous NA, Alzahrani RA, Alqurashi RM, Alharbi SS, Azhar SJ. Immediate effect of pulsed high-intensity neodymium-doped yttrium aluminum garnet (Nd: YAG) laser on staphylococcus aureus and pseudomonas aeruginosa growth: an experimental study. J Phys Ther Sci. 2019 Nov;31(11):925-930. doi: 10.1589/jpts.31.925. Epub 2019 Nov 26. PMID 31871379
- [Result] Farivar S, Malekshahabi T, Shiari R. Biological effects of low level laser therapy. J Lasers Med Sci. 2014 Spring;5(2):58-62. PMID 25653800
- [Result] Ahmad MA, A Hamid MS, Yusof A. Effects of low-level and high-intensity laser therapy as adjunctive to rehabilitation exercise on pain, stiffness and function in knee osteoarthritis: a systematic review and meta-analysis. Physiotherapy. 2022 Mar;114:85-95. doi: 10.1016/j.physio.2021.03.011. Epub 2021 Mar 26. PMID 34654554
- [Result] Roerdink RL, Dietvorst M, van der Zwaard B, van der Worp H, Zwerver J. Complications of extracorporeal shockwave therapy in plantar fasciitis: Systematic review. Int J Surg. 2017 Oct;46:133-145. doi: 10.1016/j.ijsu.2017.08.587. Epub 2017 Sep 7. PMID 28890412
- [Result] Mariotto S, de Prati AC, Cavalieri E, Amelio E, Marlinghaus E, Suzuki H. Extracorporeal shock wave therapy in inflammatory diseases: molecular mechanism that triggers anti-inflammatory action. Curr Med Chem. 2009;16(19):2366-72. doi: 10.2174/092986709788682119. PMID 19601786
- [Result] Lohrer H, Nauck T, Dorn-Lange NV, Scholl J, Vester JC. Comparison of radial versus focused extracorporeal shock waves in plantar fasciitis using functional measures. Foot Ankle Int. 2010 Jan;31(1):1-9. doi: 10.3113/FAI.2010.0001. PMID 20067715
- [Result] Melese H, Alamer A, Getie K, Nigussie F, Ayhualem S. Extracorporeal shock wave therapy on pain and foot functions in subjects with chronic plantar fasciitis: systematic review of randomized controlled trials. Disabil Rehabil. 2022 Sep;44(18):5007-5014. doi: 10.1080/09638288.2021.1928775. Epub 2021 May 26. PMID 34038642
- [Result] Diaz Lopez AM, Guzman Carrasco P. [Effectiveness of different physical therapy in conservative treatment of plantar fasciitis: systematic review]. Rev Esp Salud Publica. 2014 Jan-Feb;88(1):157-78. doi: 10.4321/S1135-57272014000100010. Spanish. PMID 24728397
- [Result] Thong-On S, Bovonsunthonchai S, Vachalathiti R, Intiravoranont W, Suwannarat S, Smith R. Effects of Strengthening and Stretching Exercises on the Temporospatial Gait Parameters in Patients With Plantar Fasciitis: A Randomized Controlled Trial. Ann Rehabil Med. 2019 Dec;43(6):662-676. doi: 10.5535/arm.2019.43.6.662. Epub 2019 Dec 31. PMID 31918529
- [Result] Jarde O, Diebold P, Havet E, Boulu G, Vernois J. Degenerative lesions of the plantar fascia: surgical treatment by fasciectomy and excision of the heel spur. A report on 38 cases. Acta Orthop Belg. 2003 Jun;69(3):267-74. PMID 12879710
- [Result] Thompson JV, Saini SS, Reb CW, Daniel JN. Diagnosis and management of plantar fasciitis. J Am Osteopath Assoc. 2014 Dec;114(12):900-6. doi: 10.7556/jaoa.2014.177. PMID 25429080